CLINICAL TRIAL: NCT00820963
Title: Randomized Study of Normal-fractionated Radiotherapy Versus Hypofractionated Radiotherapy Versus Chemotherapy in Patients Over 60 Years With Malignant Glioma
Brief Title: Standard Radiation Therapy, Higher-Dose Radiation Therapy, or Chemotherapy in Treating Older Patients With Glioblastoma Multiforme
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000626713; LEONB-ET2005-006; LEONB-Nordic Glioma Adulte; INCA-RECF0031; EUDRACT-2006-003606-25; SPRI-LEONB-ET2005-006
Record Dates: First submitted 2009-01-09; First posted 2009-01-12 (Estimated); Last update posted 2011-05-12 (Estimated); Status verified 2009-07

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult giant cell glioblastoma; adult glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma | interventions — Temozolomide; Radiotherapy

ARMS (3):
- Arm I (Experimental): Patients undergo standard radiotherapy 5 days a week for 6 weeks.
  Interventions: Radiation: radiation therapy
- Arm II (Experimental): Patients undergo hypofractionated radiotherapy 5 days a week for 2 weeks.
  Interventions: Radiation: hypofractionated radiation therapy
- Arm III (Experimental): Patients receive oral temozolomide on days 1-5. Treatment repeats every 4 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: temozolomide

INTERVENTIONS:
Drug: temozolomide — Given orally
  Arms: Arm III
Radiation: hypofractionated radiation therapy — Patients undergo hypofractionated radiotherapy
  Arms: Arm II
Radiation: radiation therapy — Patients undergo standard radiotherapy
  Arms: Arm I

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Giving radiation therapy in higher doses over a shorter period of time may kill more tumor cells and have fewer side effects. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. It is not yet known whether standard radiation therapy, higher-dose radiation therapy, or chemotherapy is more effective in treating older patients with glioblastoma multiforme.

PURPOSE: This randomized phase III trial is studying standard radiation therapy to see how well it works compared with higher-dose radiation therapy or chemotherapy in treating older patients with glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the survival of patients over 60 with glioblastoma multiforme treated with standard radiotherapy vs hypofractionated radiotherapy vs chemotherapy.

Secondary

* Compare the quality of life (QLQ-C30) of these patients.
* Compare the safety, tolerance, and toxicity of these regimens.
* Assess the pharmacoeconomic cost of these regimens.

OUTLINE: This is a multicenter study. Patients are randomized to 1 of 3 treatment arms.

* Arm I: Patients undergo standard radiotherapy 5 days a week for 6 weeks.
* Arm II: Patients undergo hypofractionated radiotherapy 5 days a week for 2 weeks.
* Arm III: Patients receive oral temozolomide on days 1-5. Treatment repeats every 4 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed glioblastoma multiforme

  * Grade 4 disease (WHO)

PATIENT CHARACTERISTICS:

* WHO performance status (PS) 0-2 (PS 3-4 allowed if secondary to a neurological physical handicap)
* Life expectancy ≥ 3 months
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 10 g/dL
* Bilirubin < 1.5 times upper limit of normal (ULN)
* Transaminases ≤ 3 times ULN
* Creatinine < 1.5 times ULN
* Able to tolerate the 3 treatment options
* No other malignancy within the past 5 years except for curatively treated basal cell or squamous cell carcinoma of the skin
* No acute or chronic severe illness that, in the investigator's opinion, contraindicates participation in the study

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy, radiotherapy, or immunotherapy
* Concurrent corticosteroids allowed provided patient is receiving the lowest dose necessary for optimal functioning

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2006-07; Primary Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Duration of survival

CONTACTS AND LOCATIONS:
Overall Officials: Didier Frappaz, MD — Centre Leon Berard
Locations (1):
- Centre Leon Berard, Lyon, France